CLINICAL TRIAL: NCT06880900
Title: Developing a Clinical Practice Guideline With The Delphi Technique for Evaluation and Counseling of Women's Sexual Health
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Handan Eriten tilaver, lecturer, Istanbul University - Cerrahpasa
Other Study IDs: HEritentilaver-IUC-PhD
Record Dates: First submitted 2024-12-29; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Female Sexual Dysfunction (FSD); Sexuality and Reproductive Issues
Keywords: female sexual dysfunction; Clinical Practice Guideline; Delphi Technique; Women's Sexual Health
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Type of Research The research will be conducted prospectively and methodologically. The Delphi Technique, one of the qualitative research methods, will be used.

Location and Time of Research Data collection will take place between April 12, 2023, and June 12, 2024, at universities, non-governmental organizations (NGOs) operating in the field of sexual health, and hospitals located in Istanbul.

Population and Sample of the Research A purposive sampling method will be used to select the participant group. Experts in sexual health working in universities, counseling centers, private and public hospitals, including nurses, physicians, psychologists, and academicians, as well as women with and without sexual dysfunction, will be included in the expert opinion team.

The ideal group size for the Delphi technique is reported to be 10-20 experts, with a minimum of 7, although this number may vary depending on the subject (Şahin, 2001). In this study, the target is to include 15 participants from each group, representing different fields, for a total of 90 participants.

Data Collection Before data collection, approval will be obtained from the Istanbul University-Cerrahpaşa Non-Interventional Clinical Research Ethics Committee and institutional permission from the Istanbul University-Cerrahpaşa, Cerrahpaşa Medical Faculty Hospital, Gynecology and Obstetrics Polyclinic.

The research will consist of two main stages. In the first stage, a clinical practice guide for evaluating and counseling women's sexual health will be created using the Delphi technique. In the second stage, the guide will be made available, and feedback will be collected from practitioners and women regarding the guide.

The Delphi technique, which will be used in the first stage, is a valid and reliable data collection method that systematically gathers expert opinions. It also allows for consensus to be reached in cases where there are differences of opinion. One of the applications of the Delphi technique is the development of standards.

Clinical Practice Guidelines are developed worldwide using three different Delphi methods: de novo, translated guides, and adaptation. In this study, the de novo Delphi method is planned to be used. The de novo guideline development method is employed when no previous guideline exists for the field of study or when existing guidelines have lost their validity. This method includes steps such as selecting the topic, forming working groups, preparing a draft guideline based on evidence and recommendations, presenting the draft to expert opinion, publishing the final guideline, delivering it to the target audience, and re-evaluating and updating it.

In this study, instead of the classical Delphi technique, the E-Delphi technique will be used with the help of electronic communication tools. The research, which will be completed after three Delphi sessions, will involve contacting participants via email and telephone.

In the first stage, experts will be identified, and face-to-face meetings will be conducted with participants for introductions. The participants' views on evaluating women's sexual health and sexual health care standards will be collected over three separate sessions using the Delphi method.

In the second stage, the guide created will be provided to healthcare workers, and it will be expected that the sexual health of women with and without sexual dysfunction will be evaluated and counseled according to this guide. Feedback from practitioners and women regarding the guide will be collected during this stage. This pilot study will be applied to 10 healthcare workers and 10 women with and without sexual dysfunction. Participants' views on the guide will be evaluated using the "Guide Satisfaction Survey (Appendix-4)."

Data Collection Tool Separate data collection tools will be used for each of the three Delphi sessions.

In the first Delphi session, the "I. Delphi Survey (Appendix-2)" will include open-ended questions addressing the research problem and demographic information. Participants will also receive the "Invitation Text (Appendix-1)" and "Informed Consent Form (Appendix-3)" containing general information about the study process and the Delphi technique.

In the second Delphi session, suggestions from the I. Delphi Survey and a literature review conducted before the sessions will be used to create standard items. These items will be compiled into a Likert-type survey, called the "II. Delphi Survey," designed to gather participants' opinions on the created items and determine their level of agreement. Participants will also be asked to add any new items, comments, or suggestions they may have.

In the third Delphi session, standard items resulting from the evaluation of data from the second Delphi session will be compiled into a Likert-type su

ELIGIBILITY:
Inclusion Criteria:

* Women with sexual dysfunction
* Women without any sexual dysfunction
* Health professionals who specialize in women's sexual health (physician, nurse/midwife, psychologist, academic)
* Women and health professionals who agree to participate in the study

Exclusion Criteria:

* Men with sexual dysfunction
* Men without any sexual dysfunction
* Healthcare professionals (physician, nurse/midwife, psychologist, academic) who do not have expertise in women's sexual health
* Women who do not agree to participate in the study and health professionals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 90
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-04-03 (Estimated); Study Completion 2025-06-03 (Estimated)

PRIMARY OUTCOMES:
I. Delphi Survey | 2 month
  In the first Delphi session, the "I. Delphi Survey (Appendix-2)" will include open-ended questions addressing the research problem and demographic information. Qualitative analyses will be conducted on the answers given to open-ended questions. Therefore, there is no cut-off value or score information in the survey study.

SECONDARY OUTCOMES:
pilot study | 5 month
  n the second stage, the guide created will be provided to healthcare workers, and it will be expected that the sexual health of women with and without sexual dysfunction will be evaluated and counseled according to this guide. Feedback from practitioners and women regarding the guide will be collected during this stage. This pilot study will be applied to 10 healthcare workers and 10 women with and without sexual dysfunction. Participants' views on the guide will be evaluated using the "Guide Satisfaction Survey (Appendix-4)."

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Üniversitesi-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No